CLINICAL TRIAL: NCT05858697
Title: Weight Development in Children With Obesity After Declining Participation in a Community-based Lifestyle Intervention.
Brief Title: Weight Development in Children With Obesity After Declining Treatment
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus County, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0367531, 2916
Record Dates: First submitted 2023-04-26; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-01

CONDITIONS: Obesity, Child
Keywords: Lifestyle intervention; refusal of treatment; effect, long term
MeSH Terms: conditions — Pediatric Obesity; Treatment Refusal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Declining group: Children with obesity 5-7 years of age who were invited to the intervention but declined participation.
  Interventions: Other: Declining participation in the Aarhus intervention
- Interventions group: Children with obesity 5-7 years of age who accepted and subsequently received treatment.
  Interventions: Behavioral: Participation in the Aarhus intervention
- 'Non intervention' group: Children with obesity at age 5-7 years living in Aarhus, who were never invited to participate in the lifestyle interventions.

INTERVENTIONS:
Other: Declining participation in the Aarhus intervention — Each year a fraction of the children invited into the Aarhus intervention decline to participated.
  Groups: Declining group
Behavioral: Participation in the Aarhus intervention — A community-based multicomponent family-centered lifestyle intervention which included visits at home and weekly supervised physical activity. The intervention has a maximum duration of one year.
  Groups: Interventions group

SUMMARY:
Childhood obesity is a major health concern and lifestyle intervention is recommended as the cornerstone in the weight loss treatment. However, only limited knowledge exists in relation to characterization and follow-up of children who decline participation in a lifestyle intervention. The aim of this study is to investigate the long-term development in BMI z-score for children with obesity who decline to participate in a lifestyle intervention.

This study identified approximately 170 children with obesity who declined treatment in a community-based lifestyle intervention. The development in BMI z-score for these children will be compared to children enrolled in the lifestyle intervention (i.e. treatment) and children who were never invited.

Data from different sources will be used to answer the research question (intervention registries, health check-ups at school and Danish registries).

DETAILED DESCRIPTION:
Childhood obesity has been associated with increased risk of poorer mental health, later non-communicable lifestyle diseases (e.g. prediabetes, sleep apnea), and of continued excess body weight into adulthood. Multi-component family-centered lifestyle intervention seems to be the cornerstone in the treatment. However, only limited knowledge exists regarding weight development in children with obesity who decline to participate in such a lifestyle intervention. The aim of this study is therefore to investigate the long-term development in BMI z-score in children with obesity from 5 to 7 years of age who declined to participate in a lifestyle intervention. The development in BMI z-score for these children will be compared to children accepting the treatment and children who were never invited. A secondary aim is to investigate the potentially modifying effects of socioeconomic status (SES).

The participants:

This cohort study will include children from the city of Aarhus with a baseline visit between January 1st 2010 and June 30th 2020 children. The inclusion criteria are 1) 5-7 years of age and 2) obesity at baseline. Obesity will be defined by the International Obesity Task Force (IOTF) as BMI ≥ 30kg/m2 for age and gender. BMI z-score will be calculated be external reference population (WHO).

The expected number of children included:

* App. 150-170 children with obesity who declined to participate in the Aarhus intervention (Declining group).
* App. 400 children with obesity accepted participation and received treatment in a multicomponent family-centered lifestyle intervention (intervention group).
* App. 700-800 children with obesity living in Aarhus, who were not invited to participate in the lifestyle intervention (Non-intervention group)

Data sources:

* Participants will be identified using data from the municipality register.
* Anthropometrical data will be extracted from TM-Sund (Aarhus). TM-Sund is a database used to store data on anthropometrics obtained at health checks by specialized school nurses, Denmark.
* Data on SES, immigration and psychiatric illness will be obtained from Danish National registries.

Statistics:

A multiple imputation (MI) with chained equations will be applied to replace missing data regarding socioeconomic status and immigration, if missing data causes the models to lose substantial amount of observations, m=100. An adjusted mixed effects model with splines will be used to describe the development in BMI z-score for children declining participation and compare those to the reference and to the intervention groups. Knots will be placed at baseline and after ½, 1, 3 and 10.5 year. The model will be adjusted for age, BMI z-score, gender, family type, highest completed household education, equalized household income, immigration status, psychiatric diagnosis and psychiatric diagnosis (parents), zip code / distance to treatment center at baseline.

Ethics & permissions:

The local health ethics committee has approved the project, including data transfer (rec.no 1-45-70-27-20).

The project is internally reported to the University of Aarhus (rec no. 2916) The project has achieved approval from The Danish Data Protection Agency and the Principal Investigator has been granted accessed to register data from Statistics Denmark.

A full plan for analytics has been completed.

ELIGIBILITY:
Inclusion Criteria:

1. 5-7 years of age
2. obesity at baseline as defined by the International Obesity Task Force (IOTF) as BMI ≥ 30kg/m2 for age and gender.

Exclusion Criteria:

1. More than 6 months between a baseline visit and the next observation with a BMI z score
2. First declining and subsequently accepting the intervention.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will include children with obesity from the city of Aarhus with a baseline visit between January 1st 2010 and June 30th 2020 children.
Sampling Method: Non-Probability Sample
Enrollment: 1273 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
The annual change in BMI z-score from baseline for children with obesity declining a lifestyle intervention and the difference in the annual change in BMI z-score compared to children in the intervention and the no-intervention group. | Baseline visit between 1st of January 2010 to 30th of June 2020.
  The annual change in BMI z-score from baseline will be modelled by using a mixed effect model with splines and be compared 1) to children accepting the treatment and 2) to children who were never invited to participate. These models will be displayed as both crude analyses and adjusted for child and parent's characteristics at baseline

SECONDARY OUTCOMES:
Different associations of the annual change in BMI z-score in subgroups (immigration and socioeconomic status) of children declining the intervention compared to children in the intervention and the no-intervention group, | Baseline visit between 1st of January 2010 to 30th of June 2020.
  A modification analysis will be applied by adding the dichotomized variables income (dichotomized by the median), education (≤12 vs ≥13 years of education) and immigration status (Danish origin vs immigrant) as interactions term to the mixed model.

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided